CLINICAL TRIAL: NCT01134835
Title: PPAR-gamma: a Novel Therapeutic Target in Asthma?
Brief Title: PPAR-gamma: a Novel Therapeutic Target for Asthma?
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: safety concerns with pioglitazone
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 08028
Record Dates: First submitted 2010-05-28; First posted 2010-06-02 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- IMP Pioglitazone (Experimental): Pioglitazone 30mg daily by mouth for 4 weeks then 45mg daily for 8 weeks and placebo 30mg daily by mouth for 4 weeks then 45mg daily for 8 weeks.
  Interventions: Drug: IMP Pioglitozone
- Placebo (Placebo Comparator): Placebo 30mg daily by mouth for 4 weeks then 45mg daily for 8 weeks and placebo 30mg daily by mouth for 4 weeks then 45mg daily for 8 weeks.
  Interventions: Other: placebo

INTERVENTIONS:
Other: placebo — placebo 30mg daily by mouth for 4 weeks then 45mg daily for 8 weeks
  Arms: Placebo
Drug: IMP Pioglitozone — Pioglitazone 30mg daily by mouth for 4 weeks then 45mg daily for 8 weeks and placebo 30mg daily by mouth for 4 weeks then 45mg daily for 8 weeks.
  Arms: IMP Pioglitazone

SUMMARY:
To test the hypothesis that stimulation of PPAR-γ receptors has a therapeutic role in the treatment of asthma.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 of either sex with a clinical diagnosis of asthma,
* FEV1 ≥ 60% predicted and an increase in FEV1 of greater than 12% following inhaled salbutamol 400μg or Peak Expiratory Flow (PEF) variability >12% during run-in.
* Allowed medication: 0-800μg inhaled beclomethasone diproprionate or equivalent and as required short acting beta agonist.

Exclusion Criteria:

* Current smoking,
* > 10 pack years smoking history,
* Treatment with leukotriene antagonists,
* Liver or cardiovascular disease,
* Oral steroid treatment or exacerbation within 6 weeks,
* Females who are pregnant, lactating or not using adequate contraception,
* Any contra-indication to pioglitazone (hypersensitivity to pioglitazone, cardiac failure, history of cardiac failure, hepatic impairment, diabetic ketoacidosis),
* Oral or insulin treatment for diabetes,
* Treatment with gemfibrozil or rifampicin.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2010-06; Primary Completion 2012-02 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
FEV1 after 12 weeks treatment | week 12

SECONDARY OUTCOMES:
Change in symptoms | 12 weeks
  Change over 12 weeks in daily asthma symptoms, mean morning and evening PEF, Juniper asthma control questionnaire and asthma quality of life questionnaire scores, exhaled nitric oxide level, bronchial hyper-responsiveness, induced sputum cell counts and analysis detailed above, adverse effects

CONTACTS AND LOCATIONS:
Locations (1):
- Nottingham University Hospitals NHS Trust, Nottingham, United Kingdom

REFERENCES:
- [Derived] Anderson JR, Mortimer K, Pang L, Smith KM, Bailey H, Hodgson DB, Shaw DE, Knox AJ, Harrison TW. Evaluation of the PPAR-gamma Agonist Pioglitazone in Mild Asthma: A Double-Blind Randomized Controlled Trial. PLoS One. 2016 Aug 25;11(8):e0160257. doi: 10.1371/journal.pone.0160257. eCollection 2016. PMID 27560168